CLINICAL TRIAL: NCT04882449
Title: Surveillance and Alert-based Multiparameter Monitoring to Reduce Worsening Heart Failure Events - SCALE-HF1
Brief Title: Surveillance and Alert-based Multiparameter Monitoring to Reduce Worsening Heart Failure Events
Acronym: SCALE-HF1
Status: Completed | Type: Observational
Sponsor: Bodyport Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00107534
Record Dates: First submitted 2021-05-06; First posted 2021-05-12 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
Keywords: Bodyport; Heart Failure; Decompensation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | US Export: No

GROUPS / COHORTS (1):
- Bodyport Cardiac Scale: All subjects will be given the Bodyport Cardiac Scale to use
  Interventions: Device: Bodyport Cardiac Scale

INTERVENTIONS:
Device: Bodyport Cardiac Scale — The Bodyport Cardiac Scale is capable of measuring key HF parameters of congestion and cardiac perfusion on a regular basis in a patient's home. These data will be combined into a composite index that may be used to identify patients at increased risk for decompensation, inform the reason for their decline, and offer the possibility to remotely optimize therapy to prevent further worsening HF.
  Other Names: Bodyport Inc.

SUMMARY:
The main goal of this study is to use data from the Bodyport Cardiac Scale to help detect of worsening heart failure (HF) early.

DETAILED DESCRIPTION:
The overarching goal of this prospective, multicenter study is to utilize data from the Bodyport Cardiac Scale to develop an index that allows for the early detection of worsening heart failure (HF). The Bodyport Cardiac Scale is capable of measuring key HF parameters of congestion and cardiac perfusion on a regular basis in a patient's home. These data will be combined into a composite index that may be used to identify patients at increased risk for decompensation, inform the reason for their decline, and offer the possibility to remotely optimize therapy to prevent further worsening HF.

The SCALE-HF program will consist of multiple phases. For SCALE-HF 1, patients will be prospectively enrolled and utilize the Bodyport Cardiac Scale on a daily basis. Patients and clinicians will be blinded to the results other than data readily available from other devices such as body weight. There will be no attempt to influence clinical practice. Patients will be followed remotely for suspected clinical events.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent before trial enrollment
2. Age ≥ 18 years
3. A diagnosis of symptomatic HF including a worsening HF event in the preceding 12 months. Worsening HF events will be determined by local clinician-investigators and will typically include the following: a) HF symptoms (eg, dyspnea, fatigue); b) HF signs (eg, elevated jugular venous pressure, peripheral edema), or laboratory/imaging evidence of HF (eg, pulmonary congestion on chest x-ray, elevated natriuretic peptide levels) during the event, and treatments targeting acute HF (eg, intravenous diuretics, vasodilators, or inotropes).

Exclusion Criteria:

1. Weight >170 kg
2. Use of chronic inotropic therapy
3. Prior heart transplant or currently listed for heart transplant
4. Current or planned left ventricular assistance device
5. Chronic kidney disease requiring chronic dialysis
6. Unknown left ventricular ejection fraction (LVEF). The LVEF should be based on the most recent local measurement using echocardiography, multigated acquisition scan, computed tomography scanning, magnetic resonance imaging, or ventricular angiography. Patients with preserved and reduced LVEF will be permitted in the study though enrollment may be capped to ensure no more than approximately 2/3 of the total enrollment includes patients with preserved or reduced LVEF.
7. Terminal illness other than HF, such as malignancy, or with a life expectancy of less than 1 year as determined by the enrolling clinician-investigator
8. Unable to participate in longitudinal follow-up including daily use of the Bodyport scale. Patients must be able to stand independently on the Bodyport scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 200-300 male and female participants in the US, 18 years of age or older, irrespective of left ventricular ejection fraction with symptomatic HF will be enrolled. Patients must be able to stand independently on the Bodyport scale.
Sampling Method: Non-Probability Sample
Enrollment: 329 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Devore, MD, Principal Investigator — Duke Clinical Research Institute
Locations (8):
- United States (8):
  - RecioMed Clinical Research Network, Inc., Boynton Beach, Florida
  - Cardiovascular Institute of Northwest Florida, Panama City, Florida
  - The Heart Center of Northeast Georgia Medical Center, Gainesville, Georgia
  - University of Kansas School of Medicine, Kansas City, Kansas
  - Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Temple University - Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - Self Regional Healthcare Research Center, Hodges, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambrosy AP, Fonarow GC, Butler J, Chioncel O, Greene SJ, Vaduganathan M, Nodari S, Lam CSP, Sato N, Shah AN, Gheorghiade M. The global health and economic burden of hospitalizations for heart failure: lessons learned from hospitalized heart failure registries. J Am Coll Cardiol. 2014 Apr 1;63(12):1123-1133. doi: 10.1016/j.jacc.2013.11.053. Epub 2014 Feb 5. PMID 24491689
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292
- [Background] Cleland JG, Charlesworth A, Lubsen J, Swedberg K, Remme WJ, Erhardt L, Di Lenarda A, Komajda M, Metra M, Torp-Pedersen C, Poole-Wilson PA; COMET Investigators. A comparison of the effects of carvedilol and metoprolol on well-being, morbidity, and mortality (the "patient journey") in patients with heart failure: a report from the Carvedilol Or Metoprolol European Trial (COMET). J Am Coll Cardiol. 2006 Apr 18;47(8):1603-11. doi: 10.1016/j.jacc.2005.11.069. Epub 2006 Mar 29. PMID 16630997
- [Background] Epstein AM, Jha AK, Orav EJ. The relationship between hospital admission rates and rehospitalizations. N Engl J Med. 2011 Dec 15;365(24):2287-95. doi: 10.1056/NEJMsa1101942. PMID 22168643
- [Background] Cowie MR, Anker SD, Cleland JGF, Felker GM, Filippatos G, Jaarsma T, Jourdain P, Knight E, Massie B, Ponikowski P, Lopez-Sendon J. Improving care for patients with acute heart failure: before, during and after hospitalization. ESC Heart Fail. 2014 Dec;1(2):110-145. doi: 10.1002/ehf2.12021. Epub 2015 Jan 21. PMID 28834628
- [Background] Soundarraj D, Singh V, Satija V, Thakur RK. Containing the Cost of Heart Failure Management: A Focus on Reducing Readmissions. Heart Fail Clin. 2017 Jan;13(1):21-28. doi: 10.1016/j.hfc.2016.07.002. PMID 27886926
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Derived] Ozonat K, Centen C, Smith S, Aydemir VB, Fudim M, DeVore AD. Bioimpedance phase angle is associated with increased heart failure hospitalization risk. Am Heart J. 2026 Feb;292:107288. doi: 10.1016/j.ahj.2025.107288. Epub 2025 Oct 7. PMID 41061788
- [Derived] Fudim M, Egolum U, Haghighat A, Kottam A, Sauer AJ, Shah H, Kumar P, Rakita V, Lopes RD, Centen C, Ozonat K, Smith S, Pandit J, DeVORE AD. Surveillance and Alert-based Multiparameter Monitoring to Reduce Worsening Heart Failure Events: Results From SCALE-HF 1. J Card Fail. 2025 Apr;31(4):661-675. doi: 10.1016/j.cardfail.2024.08.050. Epub 2024 Sep 17. PMID 39299540
- [Derived] Fudim M, Yazdi D, Egolum U, Haghighat A, Kottam A, Sauer AJ, Shah H, Kumar P, Rakita V, Centen C, Ozonat K, Smith S, DeVore AD. Use of a Cardiac Scale to Predict Heart Failure Events: Design of SCALE-HF 1. Circ Heart Fail. 2023 May;16(5):e010012. doi: 10.1161/CIRCHEARTFAILURE.122.010012. Epub 2023 May 16. PMID 37192288

RESULTS

PARTICIPANT FLOW:
Groups:
- Bodyport Scale: All subjects will be given the Bodyport scale to use
  Bodyport Scale: The Bodyport scale is capable of measuring key HF parameters of congestion and cardiac perfusion on a regular basis in a patient's home. These data will be combined into a composite index that may be used to identify patients at increased risk for decompensation, inform the reason for their decline, and offer the possibility to remotely optimize therapy to prevent further worsening HF.
Period: Overall Study
Arm/Group | Bodyport Scale
Started | 329
Completed | 329 (Enrolled participants contributed a minimum of one successful scale measurement and were included in primary outcome analysis.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bodyport Scale
Number analyzed (Participants) | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 319
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 107
  White | 210
  More than one race | 1
  Unknown or Not Reported | 8
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (8.6)
Left Ventricular Ejection Fraction [Count of Participants; unit: Participants]
  <=40% | 183
  41-49% | 25
  >=50 | 118
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Usable Worsening HF Events as Adjudicated by CEC
Description: Worsening HF will be defined as a composite of the following: urgent, unscheduled clinic or emergency department visit or hospital admission with a primary diagnosis of HF in which the patient exhibited new or worsening symptoms of HF on presentation, had objective evidence of new or worsening HF, and received initiation or intensification of treatment for HF.
Time Frame: Approximately 1 year
Measure: Number; unit: Adjudicated Events
Arm/Group | Bodyport Scale
Number analyzed (Participants) | 329
Adjudicated Events | 69

ADVERSE EVENTS:
Time Frame: Not Applicable, adverse event data were not collected for this study.
Description: As this is a non-significant risk device study with no safety endpoint, adverse events were not collected for this study. Due to no AE forms and no safety criteria in this observational study, all metrics related to AE Reporting (SAE and Other AE) are listed as 0.
  Patient outcomes were collected for the duration of follow-up (1 year), which include re-hospitalizations and patient deaths as a result of the natural worsening of patients' initial disease state.
Arm/Group | Bodyport Scale
All-Cause Mortality (participants affected / at risk) | 26/329
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04882449/Prot_000.pdf